CLINICAL TRIAL: NCT03217864
Title: Implementation of a Return Home With a Hospitalization at Home or With a Home Health Care Provider From the Services of Oncopneumology, Oncology and Hematology of University Hospital of Strasbourg: Observational, Prospective, Monocentric, Non-interventional Study. Advantages, Disadvantages, Limitations
Brief Title: Implementation of a Return Home With a Hospitalization at Home or With a Home Health Care Provider From the Services of Oncopneumology, Oncology and Hematology of University Hospital of Strasbourg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6843
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cancer
Keywords: Cancer; palliative care; hospitalization at home; home health care provider
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hospitalization at home is booming. It is designed to meet the demands of patients and their families to continue care at home. It partially solves the problem of the lack of places in the "long-term care" structures and allows to respond to a desire of the health policy to reduce the lengths of stay in the hospital. Hospitalization at home is also an alternative in the management of chronic patients. Nevertheless, at the moment a certain number of requests for hospitalization at home remain unsuccessful or their implementation is complicated. In addition, the number of home health care provider has increased significantly in recent years. According to the federation of home health care provider, the number of beneficiaries increased by 1.7% in 4 years. The home health care provider would support 1,200,000 patients per year.

The objective of the study is to analyze the factors participating in Implementation of a return home with a Hospitalization at home or a home health care provider during a return home project constructed with the patient and his / her relatives from the services of Oncology, oncology, hematology of the University Hospital of Strasbourg.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient for whom an application for Hospitalization at home or with a home health provider is initiated by the Oncology, Oncology or Hematology Department of the University Hospital of Strasbourg.

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years old for whom an application for Hospitalization at home or with a home health provider is initiated by the Oncology, Oncology or Hematology Department of of the University Hospital of Strasbourg.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Analysis of factors participating in Implementation of a return home with a Hospitalization at home or a home health care provider | 15 days after patient discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Laurent CALVEL, MD, PhD, Study Director — University Hospital, Strasbourg, France; Marie DEMEUSE, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service Soins Palliatifs, Strasbourg, France